CLINICAL TRIAL: NCT01622686
Title: PlainLanguageRx: Improving Medication Labels to Reduce Health Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PictureRx, LLC (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, M Brian Riley, Director of Research, PictureRx, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R43MD005805 (NIH); 1R43MD005805-01 (NIH)
Record Dates: First submitted 2012-06-11; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Health Behavior; Medication Adherence
Keywords: Prescription Labels; Low Health Literacy; Limited English Proficiency; Spanish
MeSH Terms: conditions — Health Behavior; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional prescription drug labels (No Intervention): Routine drug labels provided by the participating pharmacies
- Reformatted medication labels (Experimental): Prescription drug container labels that follow a new format and also include illustrations
  Interventions: Behavioral: PictureRx medication label

INTERVENTIONS:
Behavioral: PictureRx medication label — Reformatted medication labels that adhere to current best practices for label design and also include illustrations
  Arms: Reformatted medication labels

SUMMARY:
This randomized controlled trial seeks to test the effect of reformatted prescription drug container labels, compared to usual labels, on participants' understanding of their medications. The study will also assess the effect on self-efficacy and self-reported medication adherence. English and Spanish speaking patients are eligible, with a planned sample size of up to 500 adults.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old,
* Fluency in English or Spanish
* Manage their own prescription medicines, and
* Have recently filled at least 1 new prescription medication (e.g, a medicine or medication dose that they have not taken before) and have their new prescription bottle information with them.

Exclusion Criteria:

* Excludes health professionals (such as a doctor, nurse or pharmacist)
* Too ill to participate in an interview
* Do not have a telephone
* Having visual acuity worse than 20/50 via Rosenbaum Visual Acuity exam (eyechart)
* Persons picking up new medicines for others
* Inability to communicate in either Spanish or English
* Overt psychiatric illnesses, overt delirium or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Patient understanding of their medication regimen. | Approximately 7 days
  Patient understanding of the instructions for taking their medications correctly.

SECONDARY OUTCOMES:
Self-efficacy | Approximately 7 days
  Patients' confidence in being able to follow their medication regimen.
Self-reported adherence | Approximately 7 days
  Patient self-reported adherence to the medications filled.

CONTACTS AND LOCATIONS:
Overall Officials: M Brian Riley, MA, Principal Investigator — PictureRx, LLC
Locations (1):
- PictureRx, LLC (SAI Interactive), Chattanooga, Tennessee, United States